CLINICAL TRIAL: NCT05432206
Title: Randomized Double-blind Cross-over Placebo-controlled Trial to Study the Impact on Behavioral and Psychological Symptoms of Dementia of Medical Cannabinoids (CBD/THC) in Patients with Severe Dementia in Long-term Care Facilities in Geneva
Brief Title: MEDical CANnabis for Improving Symptoms During Severe DEMentia Disorders in Long-term Care Facility in Geneva
Acronym: MedCanDem
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fondation pour l'accueil et l'hébérement des personnes âgées (Other)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MedCanDem
Record Dates: First submitted 2022-06-08; First posted 2022-06-27 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Dementia with Behavioral Disturbance
Keywords: Dementia; Medical cannabis; Cannabinoids; Behavioral symptoms
MeSH Terms: conditions — Dementia; Behavioral Symptoms | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cannabis Sativa Oil first, then Placebo (Experimental): This arm will start with the active comparator for the first period and change to the placebo in the second period
  Interventions: Drug: Cannabis Sativa Oil; Drug: Placebo
- Placebo first, then Cannabis Sativa Oil (Experimental): This arm will start with the placebo for the first period and change to the active comparator in the second period
  Interventions: Drug: Cannabis Sativa Oil; Drug: Placebo

INTERVENTIONS:
Drug: Cannabis Sativa Oil — Cannabis Sativa oil standardized: 11 mg THC/g and 22 mg CBD/g.
Drug: Placebo — Hemp virgin seed oil

SUMMARY:
The behavioral and psychological symptoms of dementia affect up to 80% of long-term facilities residents with severe dementia. They seriously alter the quality of life of patients, relatives, and health professionals. Management involves correcting somatic and psychiatric factors and implementing non-drug interventions. Nevertheless, often drug treatments must be introduced with the limitations related to their effectiveness and adverse effects.

The investigators hypothesize that medical cannabinoids will improve neuropsychiatric and behavioral symptoms of patients with severe dementia.

The investigators assessed the feasibility and safety of administering a cannabis oil that contains tetrahydrocannabinol (THC) and Cannabidiol (CBD) during an initial study of about two years, observing an overall improvement, excellent tolerance to the treatment, and the possibility of reducing or even stopping other drugs.

This research project aims to study the efficacy of medical cannabis oil in improving the quality of life of dementia patients experimenting with behavioral and psychological symptoms.

DETAILED DESCRIPTION:
The study design is a placebo-controlled cross-over trial. The patients, the relatives, the health care professionals, and the study staff will be blinded.

Medical cannabis treatment is a cannabis oil that contains THC and CBD in a 1:2 ratio. The initial dose of 7 drops (2.5 mg THC and 5 mg CBD) will be gradually augmented and adjusted individually to a maximum of 56 drops (20 mg THC and 40 mg CBD) per day, divided into two administrations. Placebo is an edible oil with the same color, smell, and flavor as medical cannabis oil given with the same dosage scheme.

Patients will take medical cannabis oil for 8 weeks, in addition to their usual treatments.

The study is divided into two 8-week periods. Participants will be randomized 1:1 between cannabinoids/placebo and placebo/ cannabinoids sequences and will receive the cannabis oil during one of these periods and the placebo during the other.

Participants will observe a wash-out week between the two study periods, and a final observation week without treatment intake is planned at the end of the second period.

Rating scales to evaluate the efficacy will be assessed before treatment, after 28 days, at the end of periods, and at the end of the study. Blood pressure will be evaluated daily. Vital signs, blood formula, and the reduction or discontinuation of other drugs will be recorded periodically. In addition, the health professionals' and relatives' appraisals will be recorded at five-time points.

A blood test at the beginning and the end of each period will allow the evaluation of the potential drug-drug interactions and the pharmacokinetics of cannabinoids. The cytochromes P450 (1A2, 2B6, 2C9, 2C19, 2D6, 3A4/5) enzymatic activity will be evaluated by phenotyping after Geneva micro-cocktail intake. The therapeutic drug monitoring will be measured at a steady-state characterizing the plasma through levels of THC, its two metabolites, 11-hydroxy-tetrahydrocannabinol and free carboxy-tetrahydrocannabinol, and CBD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe dementia from different origins (Alzheimer's disease, vascular, mixed)
* Clinical Dementia Rating ≥3
* Persisting behavior problems (Neuropsychiatric Inventory [NPI] score > 10) notwithstanding optimal conventional treatment
* SARS-CoV-2 recovered for two weeks, or SARS-CoV-2 fully vaccinated
* Consent obtained from the representative in the medical field according to art 378 Swiss Civil Code (SCC)

Exclusion Criteria:

* Severe organ deficiency such as cardiac, pulmonary, hepatic, renal insufficiency, or unstable heart rhythm
* Symptomatic orthostatic hypotension
* Major changes or instability of psychotropic medication in the week preceding the study enrolment
* Having taken THC and/or CBD in the 7 days before enrolment
* Hemoglobin < 10 g/dl
* Severe kidney failure defined by cockcroft calculation <30 ml/mn
* Alanine aminotransferase and aspartate aminotransferase > 3x upper limit of normal
* Any other medical conditions that would prevent participation in the whole study protocol.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-09-29 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
Cohen-Mansfield Agitation Inventory Scale (CMAI) | 4 and 8 weeks - after 1 week washout
  Change from baseline in the Cohen-Mansfield Agitation Inventory score. Scores range from 29 to 203 - higher scores mean a worse outcome ( A total score >45 is usually regarded as clinically significant agitation).

SECONDARY OUTCOMES:
Neuropsychiatric Inventory (NPI) | 4 and 8 weeks - after 1 week wash-out
  Change from baseline in the Neuropsychiatric Inventory score. Scores range from 0 to 144 - higher scores mean a worse outcome.
Unified Parkinson disease rigidity scale (UPDRS) | 4 and 8 weeks - after 1 week wash-out
  Change from baseline in the Unified Parkinson disease rating scale (UPDRS - item 22) rigidity score. Scores range from 0 to 4 - higher scores mean a worse outcome.
Pain (Doloplus) | 4 and 8 weeks - after 1 week wash-out
  Change from baseline in the Doloplus score. Scores range from 0 to 30 - higher scores mean a worse outcome.
Daily activity | 4 and 8 weeks - after 1 week wash-out
  Change from baseline in the score evaluating the most incapacitating daily activity. Scores range 0 to 10 - higher scores mean a greater difficulty for patients.
Behavioral Trouble | 4 and 8 weeks - after 1 week wash-out
  Change from baseline in the score evaluating the most incapacitating behavioral trouble. Scores range 0 to 10 - higher scores mean a greater trouble.
Team | 4 and 8 weeks - after 1 week wash-out
  Score evaluating the team's impression of change. Scores range 1 to 7. Higher scores mean greater deterioration.
Family | 4 and 8 weeks - after 1 week wash-out
  Score evaluating the family's impression of change. Scores range 1 to 7. Higher scores mean greater deterioration.
Evolution of dosages for each patient | 4 and 8 weeks
  Dosage adjustments of medical cannabis and psychotropic drugs.
Change in enzymatic activity | 8 weeks
  Change in cytochromes P450 (1A2, 2B6, 2C9, 2C19,2D6 and 3A4/5 ) enzymatic activities using Geneva cocktail approach.
Therapeutic Drug Monitoring | 8 weeks
  Therapeutic drug monitoring of plasma concentrations of Tetrahydrocannabinol, 11-Hydroxy-tetrahydrocannabinol, 11-nor-9-carboxy-tetrahydrocannabinol, Cannabidiol.
Endocannabinoids | 8 weeks
  Evaluation of plasma levels of endocannabinoids - anandamide and 2-arachidonylglycerol.

OTHER OUTCOMES:
Blood Count 1 | 8 weeks
  Red Blood Cells, White blood cells, Platelets x1000/mm3
Blood Count 2 | 8 weeks
  Haemoglobin g/dL
Blood Count 3 | 8 weeks
  Hematocrit %
Blood Count 4 | 8 weeks
  Neutrophiles,Lymphocytes, Monocytes, Eosinophils and Basophils %
Blood pressure | through study completion, an average of 5 months
  Blood pressure measurements - systolic and diastolic mmHG.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Pautex, Prof., Principal Investigator — HUG
Locations (1):
- FAHPA, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bianchi F, Pautex S, Wampfler J, Curtin F, Daali Y, Desmeules JA, Broers B. Medical cannabinoids for painful symptoms in patients with severe dementia: a randomized, double-blind cross-over placebo-controlled trial protocol. Front Pain Res (Lausanne). 2023 May 24;4:1108832. doi: 10.3389/fpain.2023.1108832. eCollection 2023. PMID 37293434
- See also: Study Protocol — https://www.frontiersin.org/journals/pain-research/articles/10.3389/fpain.2023.1108832/full